CLINICAL TRIAL: NCT06765668
Title: Open-Label Phase 4 Study of CREXONT® (Carbidopa and Levodopa) Extended Release Capsules in Parkinson's Disease Patients
Brief Title: A Study of CREXONT (Carbidopa and Levodopa) Extended-Release Capsules in Participants With Parkinson's Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Impax Laboratories, LLC (Industry)
Collaborators: Amneal Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPX203-401-23
Record Dates: First submitted 2024-12-31; First posted 2025-01-09 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CREXONT ER (Experimental): Participants will receive CREXONT extended release (ER) capsules, orally, as guided by the Food and Drug Administration (FDA) approved prescribing Information. CREXONT ER capsules will contain Carbidopa (CD)/Levodopa (LD) 35.0 milligrams (mg)/140 mg and/or CD/LD 52.5 mg/210.0 mg and/or CD/LD 70.0 mg/280 mg and/or CD/LD 87.5 mg/350 mg. The initial CREXONT dosing regimen will be based on the FDA approved CREXONT prescribing information for dose conversion from prior oral CD-LD medications to CREXCONT. Thereafter the dosing regimen can be optimized as appropriate for the condition of each participant and guided by the FDA approved CREXONT prescribing information, in order to achieve the optimal balance of efficacy and tolerability for each participant.
  Interventions: Drug: CREXONT ER

INTERVENTIONS:
Drug: CREXONT ER — CREXONT ER capsule.
  Other Names: IPX203

SUMMARY:
The primary purpose of this study is to evaluate efficacy and safety of CREXONT under real world conditions in participants with Parkinson disease (PD).

ELIGIBILITY:
Inclusion Criteria:

1. Participants with PD consistent with the United Kingdom Parkinson's Disease Society Brain Bank Diagnostic Criteria and who are being treated with stable regimens of oral CD-LD.
2. Participants with a score of at least 20 units at Screening on the Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III total score in the "Off" state.
3. Participants with predictable "Off" periods at Screening defined by a score of 1 or 2 (Complexity of Motor Fluctuations) of the MDS-UPDRS Part IV B (Motor Fluctuations).
4. By history, for the 4 weeks (28 days) prior to Screening, the participant experiences.

   1. Daily predictable "wearing-off" episodes with periods of worsening motor symptoms.
   2. An average of at least 2.5 cumulative hours per day of "Off" time, during the hours the participant awake.
5. At Screening, the participant is able to differentiate "On" state from "Off" state as determined by at least 75 percentage (%) concordance with a trained rater (that is, investigator or qualified and certified site staff) in "On/Off" ratings for 8 ratings over a 4-hour training period. The concordance must include at least one "On" and one "Off" rating in this 4-hour training period.

   1. If the concordance is less than 75%, or if it does not include at least one "On" and one "Off" rating within the first 4-hour training period, a second 4-hour training period should be conducted with the participant before being considered for inclusion in the study.
   2. If during the second 4-hour training-period a concordance of at least 75% is also not achieved, or if it does not include at least one "On" and one "Off" rating, the participant cannot be included in the study.
6. At baseline (Visit 1), review of the 3-day PD diaries confirms the following:

   1. The participant is able to properly complete the PD diaries with valid entries. Inability to properly complete the diaries is indicated when more than 1 day of a diary is not returned or if more than 1 day of the diary is not valid (that is, more than 2 hours [4 half-hour periods] of the 24-hour diary day are missing); and
   2. The participant has an average of at least 2.5 hours per day of "Off" time, during the hours the participant is awake, over the 3 PD diary days; and
   3. The participant has at least 1.5 hours of cumulative "Off" time, during the hours the participant is awake, on each of the 3 PD diary days.
7. Participant is responsive to CD-LD therapy and currently being treated on a stable regimen of oral CD-LD for at least 4 weeks (greater than equal to [>=] 28 days) prior to baseline (Visit 1) and meets the following criteria:

   a. Daily Dose Requirements: i. All participants should be taking at least 100 mg of immediate-release (IR) CD-LD or 195 mg of Rytary for the first morning dose.

   ii. For participants taking IR CD-LD (with or without a bedtime dose of CR CD-LD):
   * Require a total daily dose of at least 300 mg of LD and a maximum total daily dose of less than equal to [<=]1200 mg LD (from IR CD-LD alone or from IR CD-LD in combination with a single daily bedtime dose of CR CD-LD).
   * The maximum individual dose allowed is 250 mg of LD.
   * The minimum individual dose should be at least 100 mg of LD. iii. For participants using a catechol-O-methyltransferase (COMT) inhibitor:
   * Require a total daily dose of at least 300 mg of LD and a maximum total daily dose of less than [<]1000 mg LD.
   * The maximum individual dose is 200 mg of LD. iv. For participants using Rytary:
   * Require a total daily dose of at least 585 mg of LD and a maximum total daily dose of <2100 mg LD.
   * The maximum individual dose is 685 mg of LD. b. Dose Frequency Requirement: i. If a participant is using IR/CR CD-LD alone or in combination with a COMT inhibitor, then the dosing frequency must be 3 to 6 times daily. ii. If a participant is using Rytary, then the dosing frequency must be 3 to 4 times daily.
8. Participant is able and willing to provide written informed consent prior to the conduct of any study-specific procedures.
9. Participant is able and willing to comply with the protocol, including completion of PD diaries, questionnaires, and available for all study visits and telephone calls.
10. Participants who have participated in prior CREXONT clinical studies are allowed to be enrolled in this Phase 4 study.

Exclusion Criteria:

1. Participant who, in the opinion of the clinical investigator, should not participate in the study based on the CREXONT Prescribing Information.
2. Participant had a prior neurosurgical treatment for PD (example, deep brain stimulation [DBS] surgery or neurosurgical ablation treatment procedures) or if such procedure is planned or anticipated prior to Visit 4 (Day 42) of the study.
3. Participant received the following within 4 weeks (<=28 days) prior to baseline (Visit 1)

   1. Any doses of a CR CD-LD apart from a single daily bedtime dose.
   2. Duopa.
   3. Nonselective monoamine oxidase inhibitor (MAOI).
   4. Rescue medication used to treat "off" episodes for example: apomorphine or inhaled LD (Inbrija®).
   5. Received any investigational drugs within 30 days or 5 times the half-life, whichever is longer, prior to baseline (Visit 1).
4. Participant who, in the opinion of the clinical investigator, should not participate in the study (example, based on clinical assessment, participant does not adequately comprehend the terminology needed to complete the PD diary and participant -reported outcomes, or any other reason).
5. Employees or family members of the investigator, or study site staff, or Sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-08-06 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in "GOOD ON" time per the Parkinson's Disease Diary to Day 42 | Baseline, Day 42
  "GOOD ON" time is derived from the 3-day Parkinson's disease (PD) diaries. For each day, "GOOD ON" time is calculated by adding the number of half-hour intervals in which either an "on time without dyskinesia" or "on time with non-troublesome dyskinesia" is checked.

SECONDARY OUTCOMES:
Change From Baseline in "OFF" time per the PD Diary to Day 42 | Baseline, Day 42
  "OFF" time is derived from the 3-day PD diaries. For each day, "OFF" time is calculated by adding the number of half-hour intervals in which the status "Off" is checked.

CONTACTS AND LOCATIONS:
Overall Officials: Hester Visser, MD, Study Director — Amneal Pharmaceuticals, LLC
Locations (27):
- United States (27):
  - Barrow Neurological Institute, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Parkinson's Research Centers of America - Orange County, Aliso Viejo, California
  - Parkinson's Research Centers of America - Palo Alto, Palo Alto, California
  - Visionary Investigators Network, Aventura, Florida
  - Parkinsons Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Univesity of Miami - Miller School of Medicine, Boca Raton, Florida
  - University of Miami, Miami, Florida
  - N1 Research LLC, Orlando, Florida
  - USF Parkinson's Disease and Movement Disorders Center, Tampa, Florida
  - Central DuPage Hospital - Movement Disorders Center, Winfield, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Quest Research Institute, Farmington Hills, Michigan
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - Parkinson's Research Centers of America - Long Island, Commack, New York
  - Atrium Health Wake Forest Baptist Adult Neurology - Janeway Tower, Winston-Salem, North Carolina
  - NeuroScience Research Center, LLC, Canton, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Movement Disorder Clinic of Oklahoma, Tulsa, Oklahoma
  - Neurology Consultants of Dallas, PA, Dallas, Texas
  - Texas Movement Disorder Specialists, PLLC, Georgetown, Texas
  - Icahn School of Medicine at Mount Sinai, Houston, Texas
  - The University of Texas Health Science Center at Houston- McGovern Medical School, Houston, Texas
  - Inova Neurology, Fairfax, Virginia
  - VCU Parkinsons Disease and Movement Disorders Center, Henrico, Virginia
  - MedStar Georgetown University Hospital Department of Neurology, McLean, Virginia

IPD SHARING:
Plan to Share IPD: No